CLINICAL TRIAL: NCT05142085
Title: Effect of Nano-PSO in Patients With Parkinson's Disease: Clinical Efficacy and Results in Molecular Imaging.
Brief Title: Efficacy of Nano-PSO in Parkinson's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Distribuidora Biolife SA de CV (Industry)
Responsible Party: Principal Investigator, Marie-Catherine Boll, MD,PhD, Distribuidora Biolife SA de CV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INNN0121
Record Dates: First submitted 2021-11-05; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson´s disease; punicic acid; neuroprotection; molecular imaging
MeSH Terms: conditions — Parkinson Disease | interventions — Nano-PSO

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatments are made in an independent laboratory that has a white area for packaging the placebos and the treatments with a label that is kept in a database on this site and, in its printed version, in another center.
  Boxes are prepared with a content of 5 treatments (2 placebos for 3 active ingredients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy of nano-PSO on motor and non-motors symptoms of Parkinson´s disease. (Experimental): It is the clinical trial itself where more than 140 subjects will be included:
  84 under active treatment and 56 under placebo
  Interventions: Dietary Supplement: nano-PSO; Other: placebo
- Effect of nano-PSO on molecular images of PD patients (Experimental): In this group, the study implicates performing a multitracer PET-scan before treatment, and at 6 months, to 25 subjects in the clinical trial : 15 under active treatment and 10 in the placebo group.
  Interventions: Dietary Supplement: nano-PSO; Other: placebo

INTERVENTIONS:
Dietary Supplement: nano-PSO — This active treatment will be delivered to 3 out of 5 patients
  Other Names: nanodroplet formulation of pomegranate seed oil (PSO)
Other: placebo — This treatment will be assigned to 2 out of 5 patients
  Other Names: capsules of neutral mineral oil

SUMMARY:
The present research aims to carry out a double-blind, placebo-controlled clinical trial to study the efficacy of a new antioxidant. The primary outcome variables will be the changes observed in PD-motor and non-motor symptoms scales, as well as quality of life during a 6-months period. Global impression on the treatment will be rated after this period. Likewise, presynaptic changes will be studied in positron emission tomography studies, using 2 radiotracers and a dynamic image processing in patients with Parkinson's disease.

125 patients who have a definite diagnosis of PD will be included; 25 of them will be subjected to a triple-blind, clinical and molecular study. In addition, 25 other subjects from the same Institution and from 4 other collaborating centers will be part of the clinical arm of this study during the period September 2021- September 2022.

During the first visit, various clinical data of the participants will be recorded such as: age, gender, family history, current medical conditions, and drugs dosage in addition to a comprehensive neurological examination. Subsequently, the signing of the informed consent will be obtained, and general laboratory tests and a brain RMI in 3dT1 and SWI sequences will be performed. A series of disease-specific scales will be applied in order to assess motor functional capacity, cognition, sleep, and other non-motor symptoms before drug delivery.

Randomization will be made in blocks of 5 treatments: 3 nano-PSO and 2 placebos. Treatments will be delivered in form of bottles containing 100 capsules each after baseline and intermediate visit.

25 patients will also give their consent to perform 2 PET studies (positron emission tomography) to assess presynaptic dopaminergic function. This implies conducting these studies on 2 occasions (at the beginning and at the end of treatment), with emphasis on striatal activity to study the effect of treatment with Nano-PSO.

DETAILED DESCRIPTION:
A new fatty acid extracted from the pomegranate showed unexpectedly beneficial properties after nanotechnological processing. Encouraging effects of the new substance called nano-PSO led to design the present investigation. Indeed, the substance is responsible for slowing down cognitive deterioration in Alzheimer disease models, with an evident protective mechanism against oxidative mitochondrial damage and also for increasing survival in Creutzfeldt-Jakob disease models, among other results in preclinical research. Recently, a trial realized in multiple sclerosis patients showed beneficial effects on functional outcomes. In addition, another study showed significant positive results in tyrosine-hydroxylase activity, mitochondrial enhancement, and motor function in animal models of PD under nano-PSO treatment.

Therefore, the design of a clinical trial involving 3 neurological referral centers is necessary to be able to select and include an appropriate sample of PD patients to evaluate the benefits of nano-PSO. The time of the study is limited to one year, since this treatment is already approved for commercialization as a nutritional supplement.

The first 25 included patients who also give their consent to carry out the PET study (positron emission tomography on two occasions (at the beginning and at the end of treatment), with emphasis on striatal presynaptic activity, will provide molecular hard data for evaluating efficacy of the treatment. Molecular imaging tools are evolving and nowaday able to obtain changes in dynamic and sensitive variables for the detection of changes due to treatment; also, it can correlate clinimetric and functional data with unprecedented accuracy and resolution. Post processing molecular images of involved subjects with appropriate softwares will return a series of variables including VOI analysis, general kinetic modeling, pixel-wise modeling, images in 3D and in motion, especial quantitative data processing.

After confirmation of the diagnosis and review of the criteria, the process for obtaining informed consent is carried out. An extended informed consent form was performed for the PET group of volunteers as they need during the first week of their participation a structural MRI, the FDG PET-scan and another day to perform the 18 -fluorodopa PET-scan. These studies are intended to merge images, to study the cerebral metabolism of glucose, dopamine tracing, and to process dynamic events with a P-Mode software. Patients are aware of the need to perform a second similar study after 6 months of treatment. The rest of the protocol is similar for the group subjected to the PET study n=25) and the exclusively clinical study group (n=100). It consists of the collection of elements of the medical history, blood samples analysis, ECG, and MRI review ,quality of life and Montreal Cognitive Assessment, MDS-UPDRS** , Non motor symptoms scale, PD sleep scale, H&Y stage.

The clinimetric protocol will be applied at least three times: at baseline, 3-months- after 6 months of treatment. During each interval, a questionnaire will be carried out via telephone, videoconference or video-call.

Enrolled patients will be connected constantly with a clinician through a smartphone activated only for research needs. (schedule, report of adverse events, request transportation etc. ) The protocol has been registered this year, and approved by three institutional committees: the scientific committee, the ethics and the biosafety committee. In the two other participating centers, only approval by the Research Ethics committee is required since PET-scan will not be performed in the study frame.

Molecular biomarkers:

A sample of 25 patients who firme a special informed consent will be followed with a multitracer positron emission tomography (PET) at the basal state and after 6 months of treatment. PET is an imaging technique using radiotracers to obtain functional images of the central nervous system. Neuronal loss occurs in a caudal to rostral fashion in PD, from the brainstem where the hallmark pathology still relies on the Lewy bodies in the SNc. The latter corresponds to intra-cytoplasmatic alpha-synuclein-positive staining inclusions.

Firstly, 18 F-FDG is a glucose analogue and direct marker for GLUT-1 cell membrane expression and function. This tracer allows diagnosis and differential diagnosis of PD and parkinsonian syndromes. PD is characterized by an increased uptake of FDG in striatal and thalamic areas, in comparison with cortical and cerebellar regions. This increased uptake is mostly contralateral to the most affected side. In multiple system atrophy ( MSA) a decreased uptake is seen and in the MSA-C form, with cerebellar hypometabolism.

In PD the mean annual rate of decline in FD uptake reportedly ranges from 8% to 12% in the putamen and 4-6% in the caudate, while annual decline in healthy volunteers is 0.5% and 0.7%, respectively. Autopsy studies have shown a 45% decrease in nigral cell counts during the first 10 years of PD. PET scan using 6-[ 18 F]-fluoro-L-3,4-dihydroxyphenylananine ( 18 F-FDOPA) allow quantification of striatal DOPA decarboxylase activity and storage capacity of 18 F-dopamine . This study can evaluate unlimited depth penetration and take whole body imaging despite is an expensive exam. Spatial resolution can be co-registered with structural data from MR images to provide additional anatomical context to the functional PET data. The first data analysis is both visually and quantitatively. Further dynamic data will be given by a study of striatal decarboxylase activity and storage of fluoroDOPA by the mean of a P-mode software.

Statistics Sample size was calculated to compare the primary clinical outcomes of a nano-PSO treated group of 60 to 75 subjects with a placebo group of 40 to 50 subjects. A difference of 5 points of changes in the motor scale is arbitrary expected. To estimate the distribution of this variable (changes in the MDS-UPDRS motor scale, in a sample of 16 patients recently attended allowed the calculation of a mean of 9.9 points and the standard deviation of 6.69. Assuming that those in the placebo group do not change their score, while those treated with nano-PSO earn five points, a sample of 30 subjects in each group was calculated.

Sample size calculation for the clinical essay was based on the hypothesis of a gain of 5 points in the MDS-UPDRS motor score in the treated group, assuming a placebo effect of 2 points, a mean change of 5 in the treated group. Standard deviation of 10 obtained in definite PD cases. With a value for desired power of 80% and an alpha error of 0.05, the sample size for a one-sided test of hypothesis is of 50 cases in each group. An interim analysis is planned in septembre 2022 when 30 to 50 subjects will finish the trial.

The other primary outcome is the gain in non-motor symptoms scale (NMSS) with a similar measurement.

** MDS-UPDRS motor sub scale (part III) is assessed in patients submitted to the PET study in OFF state , and further in ON of Levodopa. All the other subjects are called to come in their best ON stage during their evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Parkinson's disease confirmed with UKPDSBB and MDS clinical criteria.
* who signed the informed consent to follow the study protocol.
* Age at onset of PD: 45-60 years.
* Age at enrollment: 45-65 years
* Disease of 2 to 8 years of evolution
* Without uncontrolled chronic degenerative disease (High blood pressure, AF, dyslipidemia).
* Without uncontrolled diabetes mellitus
* With a fixed treatment during the last 3 months and throughout the study.
* A patient who does not suffer from another neurodegenerative disease.
* No symptomatic brain injury.
* A patient who can lie on his back for at least 2 hours in the OFF state of levodopa.

Exclusion Criteria:

* Patients unable to give their informed consent
* Subjects who are not able to fill out a questionnaire or cooperate during the study
* Diabetic people
* or with another uncontrolled chronic disease
* or with brain injury.

Ages: 48 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-01-03 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in MDS-UPDRS motor scale | 6 months
  The Unified PD rating scale (UPDRS) reviewed by the Movement Disorders Society is a 4 domains instrument that measures 1.- non-motor aspects of experiences of daily living ( 13 items),2.- Daily life activities (13 items). 3.- Motor examination (33 items) 4.- motor complications (6 items) Each item is scored from 0 to 4 , with the highest being the worst.
Changes in NMSS ( non-motor symptoms scale) | 6 months
  This is a scale of 8 domains (cardiovascular, sleep/fatigue, mood/cognition, vision/hallucinations atention, gastrointestinal, urinary, sexual and others. where the presence, severity and frequency are multiplied, obtaining 0 for the best score, and 360 points for the worst case.

SECONDARY OUTCOMES:
Changes in PDQ-8 | 6 months
  changes in quality of life are measured with this 8 domains scale . It is measured as a percentage, with 100% being the greatest loss of quality of life.
Modification of LEDD ( levodopa equivalent daily dose.) | 6 months
  Measured in mg) ( may be modified during the follow-up) captured as increased, unchanged or decrease) it could be reduced under the experimental treatment.
Global impression of the treatment | ...after 6 months
  This outcome is measured with an analog scale at the end of the test. (range 0-10) 10 is the best score.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Kerik Rotenberg, MD, Study Chair — INNN-MVS Department of Nuclear Medicine; Marie-Catherine Boll, MD,PhD, Principal Investigator — Clinical Research Laboratory Instituto Nacional de Neurología y Neurocirugía MVS. MEXICO CITY; Ulises Rodríguez Ortiz, MDS, Study Chair — Médica Sur Mexico
Locations (1):
- Instituto Nacional de Neurología y Neurocirugía, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Access to patients study files is authorized only to study researchers. When incorporating PI from other centers, the REDCap platform will be used.

REFERENCES:
- [Background] Chondrogiannis S, Marzola MC, Al-Nahhas A, Venkatanarayana TD, Mazza A, Opocher G, Rubello D. Normal biodistribution pattern and physiologic variants of 18F-DOPA PET imaging. Nucl Med Commun. 2013 Dec;34(12):1141-9. doi: 10.1097/MNM.0000000000000008. PMID 24128899
- [Background] Kumakura Y, Gjedde A, Danielsen EH, Christensen S, Cumming P. Dopamine storage capacity in caudate and putamen of patients with early Parkinson's disease: correlation with asymmetry of motor symptoms. J Cereb Blood Flow Metab. 2006 Mar;26(3):358-70. doi: 10.1038/sj.jcbfm.9600202. PMID 16079784
- [Background] Nanni C, Fanti S, Rubello D. 18F-DOPA PET and PET/CT. J Nucl Med. 2007 Oct;48(10):1577-9. doi: 10.2967/jnumed.107.041947. No abstract available. PMID 17909255
- [Background] Binyamin O, Larush L, Frid K, Keller G, Friedman-Levi Y, Ovadia H, Abramsky O, Magdassi S, Gabizon R. Treatment of a multiple sclerosis animal model by a novel nanodrop formulation of a natural antioxidant. Int J Nanomedicine. 2015 Nov 20;10:7165-74. doi: 10.2147/IJN.S92704. eCollection 2015. PMID 26648720
- [Background] Binyamin O, Nitzan K, Frid K, Ungar Y, Rosenmann H, Gabizon R. Brain targeting of 9c,11t-Conjugated Linoleic Acid, a natural calpain inhibitor, preserves memory and reduces Abeta and P25 accumulation in 5XFAD mice. Sci Rep. 2019 Dec 5;9(1):18437. doi: 10.1038/s41598-019-54971-9. PMID 31804596
- [Background] Binyamin O, Keller G, Frid K, Larush L, Magdassi S, Gabizon R. Continues administration of Nano-PSO significantly increased survival of genetic CJD mice. Neurobiol Dis. 2017 Dec;108:140-147. doi: 10.1016/j.nbd.2017.08.012. Epub 2017 Aug 25. PMID 28847567
- [Background] Keller G, Binyamin O, Frid K, Saada A, Gabizon R. Mitochondrial dysfunction in preclinical genetic prion disease: A target for preventive treatment? Neurobiol Dis. 2019 Apr;124:57-66. doi: 10.1016/j.nbd.2018.11.003. Epub 2018 Nov 10. PMID 30423473
- [Background] Zamora-Lopez K, Noriega LG, Estanes-Hernandez A, Escalona-Nandez I, Tobon-Cornejo S, Tovar AR, Barbero-Becerra V, Perez-Monter C. Punica granatum L.-derived omega-5 nanoemulsion improves hepatic steatosis in mice fed a high fat diet by increasing fatty acid utilization in hepatocytes. Sci Rep. 2020 Sep 17;10(1):15229. doi: 10.1038/s41598-020-71878-y. PMID 32943651
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Eidelberg D, Moeller JR, Dhawan V, Sidtis JJ, Ginos JZ, Strother SC, Cedarbaum J, Greene P, Fahn S, Rottenberg DA. The metabolic anatomy of Parkinson's disease: complementary [18F]fluorodeoxyglucose and [18F]fluorodopa positron emission tomographic studies. Mov Disord. 1990;5(3):203-13. doi: 10.1002/mds.870050304. PMID 2117706
- [Background] Eshuis SA, Maguire RP, Leenders KL, Jonkman S, Jager PL. Comparison of FP-CIT SPECT with F-DOPA PET in patients with de novo and advanced Parkinson's disease. Eur J Nucl Med Mol Imaging. 2006 Feb;33(2):200-9. doi: 10.1007/s00259-005-1904-y. Epub 2005 Oct 15. PMID 16228235
- [Background] Pysz MA, Gambhir SS, Willmann JK. Molecular imaging: current status and emerging strategies. Clin Radiol. 2010 Jul;65(7):500-16. doi: 10.1016/j.crad.2010.03.011. PMID 20541650